CLINICAL TRIAL: NCT02628626
Title: A Placebo Controlled Study of Colesevelam in Fecal Incontinence
Brief Title: A Study of Colesevelam in Fecal Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Adil Bharucha, MBBS, MD, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-005986; R01DK078924 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Fecal Incontinence; Bile Acid Malabsorption
Keywords: Incontinence; Diarrhea; Bile acid; Microbiome
MeSH Terms: conditions — Fecal Incontinence; Diarrhea | interventions — Colesevelam Hydrochloride; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in this arm will receive placebo for 4 weeks.
  Interventions: Other: Placebo
- Colesevelam and Clonidine (Active Comparator): Participants in this arm will receive a combination of colesevelam (1.875 gm twice daily) and clonidine (0.1 mg oral twice daily) for 4 weeks.
  Interventions: Drug: Colesevelam; Drug: Clonidine

INTERVENTIONS:
Drug: Colesevelam — Participants who satisfy symptom criteria in Phase 2 will be randomized in a 1:1 ratio to receive either a combination of colesevelam (1.875 gm twice daily) and clonidine (0.1 mg oral twice daily) or an identical placebo for 4 weeks.
  Other Names: Welchol
  Arms: Colesevelam and Clonidine
Drug: Clonidine — Participants who satisfy symptom criteria in Phase 2 will be randomized in a 1:1 ratio to receive either a combination of colesevelam (1.875 gm twice daily) and clonidine (0.1 mg oral twice daily) or an identical placebo for 4 weeks.
  Other Names: Catapres
  Arms: Colesevelam and Clonidine
Other: Placebo — Placebo will be identical in appearance to the active drug.
  Arms: Placebo

SUMMARY:
Compare the effects of a combination of colesevelam and clonidine to placebo on bowel symptoms in patients with urge or combined type of FI.

DETAILED DESCRIPTION:
Fecal incontinence (FI) is a common symptom that can significantly impair quality of life. There is very limited, mostly uncontrolled, evidence to support the approaches currently used to manage FI. The alpha-2 adrenergic agonist clonidine decreased the frequency of loose stools in FI patients with diarrhea. Among patients with diarrhea, clonidine decreased the proportion of days with FI; however results were not statistically significant. Uncontrolled studies suggest that the bile acid binding resin colesevelam also increased stool consistency in patients with functional diarrhea. In this study, the investigators propose to compare the effects of a combination of colesevelam and clonidine to placebo on bowel symptoms in patients with urge or combined type of FI.

ELIGIBILITY:
A. Phase 1

Inclusion Criteria:

i) Females aged 18-80 years with urge predominant or combined (i.e. urge plus passive) FI, as defined by a validated questionnaire, for at least 1 year duration will be eligible to participate.

Exclusion Criteria:

(i) History of clinically serious cardiovascular or pulmonary disease or EKG showing 2nd degree atrioventricular block or higher.

(ii) Current or past history of rectal cancer, scleroderma, inflammatory bowel disease, small bowel obstruction, congenital anorectal abnormalities, Grade 2 rectal prolapse, history of rectal resection or pelvic irradiation (iii) Neurological disorders - Spinal cord injuries, dementia (Mini-Mental status score <21), multiple sclerosis, Parkinson's disease, peripheral neuropathy (iv) Conditions precluding safe use of clonidine, i.e., symptomatic hypotension, or systolic blood pressure of <100 mm Hg on initial visit in Phase 1 of study (v) Currently pregnant or nursing women (vi) Prior history of intolerance to clonidine or colesevelam (vii) Medications Absolute - opioid analgesics. Relative - other antihypertensive agents (i.e. if there is concern about synergistic effects and hypotension). Patients using drugs with anticholinergic effects will be excluded if they are used at high doses (e.g. nortriptyline greater than 50 mg/day or amitriptyline greater than 25 mg/day). Patients who use lower doses will be eligible to participate provided the dose will be stable during the study

B. Phase 2

Inclusion Criteria:

i) Females aged 18-80 years with urge predominant or combined (i.e. urge plus passive) FI for at least 1 year, as defined by questionnaire

Exclusion criteria:

(i) Positive urine pregnancy screen

C. Phase 3

Inclusion criteria:

(i) Completion of at least 5 out of 7 days of the diary in the preceding week and 10 out of 14 in the preceding 2 weeks (ii) At least 1 episode of FI per week averaged over 2 weeks (iii) Average Bristol stool score of 3 or higher (iv) Average stool frequency of ≥1/day

Exclusion criteria (if at least one is satisfied):

(i) Missing data in bowel diaries, i.e. if patient did not record bowel symptoms data for more than 2 days in 1 week or 4 days over 2 weeks (ii) Greater than 6 liquid [Bristol 6 or 7]) stools daily (iii) Average of less than 1 bowel movement daily (iv) Average Bristol stool score <3 as assessed from analysis of bowel diaries

D. Phase 4

Inclusion criteria:

(i) All patients who complete at least 1 week of treatment with study drugs or placebo

Exclusion criteria:

(i) Patients who completed less than 1 week of treatment with study drugs or placebo

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-11; Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty-eight (88) participants were enrolled but thirty-two (32) withdrew from the study before beginning any study procedures.
Period: Overall Study
Arm/Group | Placebo | Colesevelam and Clonidine
Started | 32 | 24
Completed | 30 | 22
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Colesevelam and Clonidine | Total
Number analyzed (Participants) | 32 | 24 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (26) | 53 (29) | 50 (27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 24 | 56
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 24 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 24 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Report a 50% or Greater Reduction in Weekly Fecal Incontinence (FI) Episodes
Description: The number of participants that report a 50% or greater reduction in weekly incontinent episodes as measured by self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
Participants | 17 | 13
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.85, ANCOVA

2. Secondary Outcome: Daily Stool Frequency
Description: The number of bowel movements daily measured by self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: bowel movements per day
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
bowel movements per day | 2.4 (2.3) | 2.1 (2.0)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Approximately 4 weeks; Test type: Superiority; p = 0.24, ANCOVA

3. Secondary Outcome: Stool Consistency
Description: Stool consistency as measured by self-reported bowel diaries. Expressed in terms of the Bristol Stool Form Scale, where: 1= separate hard lumps; 2= lumpy sausage-shape; 3= cracked sausage; 4= smooth and soft sausage; 5=soft blobs; 6=mushy, fluffy pieces; 7= watery, no solid pieces.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
score on a scale | 4.1 (1.9) | 3.2 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Approximately 4 weeks; Test type: Superiority; p = 0.44, ANCOVA

4. Secondary Outcome: Number of Semi-Formed Stools Per Week
Description: The number of stools per week measured by self-reported bowel diaries where the Bristol stool score was 5, 6, or 7. (5=soft blobs; 6=mushy, fluffy pieces; 7= watery, no solid pieces)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: number of stools per week
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
number of stools per week | 1.0 (0.7) | 1.2 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.35, ANCOVA

5. Secondary Outcome: Delay of Bowel Movement
Description: The time in minutes a bowel movement can be delayed after sense of urgency to defecate as measured by self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
minutes | 2.8 (7.8) | 3.6 (8.4)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Approximately 4 weeks; Test type: Superiority; p = 0.56, ANCOVA

6. Secondary Outcome: Total Fecal Incontinence Episodes
Description: The total number of fecal incontinence episodes per week as measured by self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: incontinence episodes per week
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
incontinence episodes per week | 4.2 (4.4) | 4.8 (3.7)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.55, ANCOVA

7. Secondary Outcome: Volume of Fecal Incontinence
Description: The volume of fecal incontinence measured as the number of incontinent episodes per week as categorized by small (staining only), moderate (requiring change of underwear) or large (requiring change of all clothes) in self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: incontinent episodes per week
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
incontinent episodes per week
  Small (staining only) | 2.4 (1.8) | 3.3 (3.0)
  Moderate (requires change of underwear) | 0.9 (1.7) | 2.0 (2.6)
  Large (requires complete change of clothes | 1.3 (2.2) | 2.4 (6.2)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Small (staining only); Test type: Superiority; p = 0.11, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Colesevelam and Clonidine; Moderate (requires change of underwear); Test type: Superiority; p = 0.06, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Colesevelam and Clonidine; Large (requires complete change of clothes); Test type: Superiority; p = 0.36, ANCOVA

8. Secondary Outcome: Percent of Incontinent Bowel Movements Pre-treatment
Description: The percentage of bowel movements that were incontinent prior to treatment initiation, per self-reported bowel diaries.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percent of incontinent bowel movements
Units Other Than Participants: Bowel Movements
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
Number analyzed (Bowel Movements) | 1362 | 1013
percent of incontinent bowel movements | 45 (9) | 40 (10)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.18, ANCOVA

9. Secondary Outcome: Percent of Incontinent Bowel Movements During Treatment
Description: The percentage of bowel movements that were incontinent during treatment, per self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent of incontinent bowel movements
Units Other Than Participants: Bowel Movements
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
Number analyzed (Bowel Movements) | 1419 | 1086
percent of incontinent bowel movements | 27 (8) | 28 (9)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.04, ANCOVA

10. Secondary Outcome: Percent of Incontinent Bowel Movements to be Semi-Formed Stools Pre-Treatment
Description: The percentage of incontinent bowel movements where the Bristol stool score was 5, 6 or 7. (5=soft blobs; 6=mushy, fluffy pieces; 7= watery, no solid pieces), pre-treatment, per self-reported bowel diaries.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percent of semi-formed stools
Units Other Than Participants: Incontinent Bowel Movements
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
Number analyzed (Incontinent Bowel Movements) | 613 | 405
percent of semi-formed stools | 61 (8) | 76 (8)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.29, ANCOVA

11. Secondary Outcome: Percent of Incontinent Bowel Movements to be Semi-Formed Stools During Treatment
Description: The percentage of incontinent bowel movements where the Bristol stool score was 5, 6 or 7. (5=soft blobs; 6=mushy, fluffy pieces; 7= watery, no solid pieces) during treatment, per self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent of semi-formed stools
Units Other Than Participants: Incontinent Bowel Movements
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
Number analyzed (Incontinent Bowel Movements) | 383 | 304
percent of semi-formed stools | 67 (8) | 61 (10)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.39, ANCOVA

12. Secondary Outcome: Severity of Bowel Symptoms
Description: The Fecal Incontinence Symptom Severity (FISS) score is based on five questions; (1) the frequency of FI; (2) the type of FI (stool only, liquid or mucus only, both liquid/mucus and stool, or gas only); (3) the amount of stool leaked (small, moderate, or large); (4) the frequency of having to rush to the toilet; and (5) the frequency of having stool leak without warning. Questions 4 & 5 are merged to determine if the participant has passive FI (FI without warning), urge FI, both, or neither. The responses to the questions are assigned physician-derived weights and added together for a total score of 4 to 13. The higher the score the more severe the FI symptoms.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
score on a scale | 6 (3.2) | 4.6 (3.6)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority; p = 0.07, ANCOVA

13. Secondary Outcome: Severity of Fecal Incontinence
Description: Measured by the Fecal Incontinence Severity Index (FISI). It is a validated 4-item scale used to assess the frequency (never, 1-3 times a month, once a week, 2 or more times per week but not daily, once a day, 2 or more times per day) of 4 different types of FI (gas, mucus, liquid stool, solid stool). Each of the four types of FI is awarded a number of points, depending on the frequency at which that type of incontinence is experienced. The points are totaled and the scores can range from 0 to 61, where the higher the score, the higher the perceived severity of the fecal incontinence.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
score on a scale | 28 (15) | 22 (18)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Test type: Superiority — approximately 4 weeks post-treatment; p = 0.12, ANCOVA

14. Secondary Outcome: Fecal Incontinence Quality of Life (FI-QoL)
Description: The Fecal Incontinence Quality of Life questionnaire measures specific quality of life issues expected to affect patients with fecal incontinence. The questions are grouped into four categories: lifestyle (10 questions), coping (9 questions), depression (7 questions), and embarrassment (3 questions). Each category is scored from 1 to 4. The scale scores are calculated by adding the numerical values of all responses in that specific scale and then dividing by its number of items. Higher scores indicate a better quality of life.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
score on a scale
  Lifestyle score | 2.7 (0.9) | 2.7 (0.9)
  Coping score | 2.0 (0.6) | 2.1 (0.8)
  Depression Score | 3.1 (0.6) | 3.1 (0.8)
  Embarrassment score | 2.6 (0.9) | 2.5 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Lifestyle Score; Test type: Superiority; p = 0.67, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Colesevelam and Clonidine; Coping Score; Test type: Superiority; p = 0.80, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Colesevelam and Clonidine; Depression Score; Test type: Superiority; p = 0.49, ANCOVA
Statistical Analysis 4: Comparison: Placebo vs Colesevelam and Clonidine; Embarrassment Score; Test type: Superiority; p = 0.60, ANCOVA

15. Secondary Outcome: Loperamide Tablets Per Week
Description: The number of tablets of loperamide used, per self-reported bowel diaries.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: tablets per week
Arm/Group | Placebo | Colesevelam and Clonidine
Number analyzed (Participants) | 30 | 22
tablets per week | 1.9 (2) | 6 (5)
Statistical Analysis 1: Comparison: Placebo vs Colesevelam and Clonidine; Approximately 4 weeks post-treatment; Test type: Superiority; p = 0.78, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to the end of study participation, for a total of approximately 12 weeks on each participant.
Arm/Group | Placebo | Colesevelam and Clonidine
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/24
Other Adverse Events (participants affected / at risk) | 4/32 | 6/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Colesevelam and Clonidine (N=24)
Nausea and bloating (General disorders) | 0 (0) | 2 (2)
Intercurrent Illness (General disorders) | 1 (1) | 2 (2)
Difficulty swallowing pills (General disorders) | 2 (2) | 2 (2)
Insomnia (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT02628626/Prot_SAP_000.pdf